CLINICAL TRIAL: NCT02731833
Title: A Clinical Study Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Brief Title: Short Term Clinical Study Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205710
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Test dentifrice (Experimental): Participants will be instructed to dose a dry toothbrush with a full strip (1 inch) of toothpaste. Participants will then brush each of the two selected sensitive test teeth first followed by the whole mouth thoroughly for at least 1 minute
  Interventions: Other: stannous fluoride
- Control dentifrice (Active Comparator): Participants will be instructed to dose a dry toothbrush with a full strip (1 inch) of toothpaste. Participants will then brush whole mouth thoroughly for at least 1 minute
  Interventions: Other: sodium monofluorophosphate

INTERVENTIONS:
Other: stannous fluoride — 0.454% weight by weight (w/w) stannous fluoride containing 1100ppm fluoride
  Arms: Test dentifrice
Other: sodium monofluorophosphate — 0.76% w/w sodium monofluorophosphate containing 1000ppm fluoride
  Arms: Control dentifrice

SUMMARY:
This single centre, comparative design study will be used to investigate the efficacy of an experimental stannous fluoride containing dentifrice in relieving dentinal hypersensitivity (DH) after short term use compared with a standard fluoride dentifrice

DETAILED DESCRIPTION:
This will be a single centre, three day, randomised, examiner blind, two treatment arm, parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected test teeth), controlled study, in participants with at least two sensitive teeth that meet all the criteria at the screening and baseline (pre-treatment) visits. Dentinal hypersensitivity will be assessed at baseline (pre-treatment), post-treatment and after 3 days twice daily brushing

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Aged 18-65 years inclusive
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: a) No clinically significant and relevant abnormalities of medical history or oral examination. b) Absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements
* Self-reported history of dentinal hypersensitivity (DH) lasting more than six months but not more than 10 years
* Minimum of 20 natural teeth
* Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria: Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR), Tooth with MGI score =0 adjacent to the test area (exposed dentine) only [Lobene, 1986] and a clinical mobility of ≤1, Tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response)
* Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), that meet all of the following criteria: Tooth with signs of sensitivity, measured by qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff sensitivity score ≥ 2)

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study
* Recent history (within the last year) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes or Any condition which, in the opinion of the investigator, causes xerostomia
* Dental prophylaxis within 4 weeks of Screening or Tongue or lip piercing or presence of dental implants
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening and teeth bleaching within 8 weeks of Screening
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine
* Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening (participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients)
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs
* Currently taking antibiotics or has taken antibiotics within 2 weeks of Baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2016-04-01; Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mississauga, Ontario, Canada

REFERENCES:
- [Derived] Creeth J, Gallob J, Sufi F, Qaqish J, Gomez-Pereira P, Budhawant C, Goyal C. Randomised clinical studies investigating immediate and short-term efficacy of an occluding toothpaste in providing dentine hypersensitivity relief. BMC Oral Health. 2019 Jun 4;19(1):98. doi: 10.1186/s12903-019-0781-x. PMID 31164116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at single clinical site in Canada.
Pre-assignment Details: A total of 229 participants were screened. Out of which 222 participants were randomized. 7 participants were not randomized because these participants did not meet study criteria.
Groups:
- Stannous Fluoride: Participants were instructed to dose a dry toothbrush with a full strip (1 inch) of experimental dentifrice containing 0.454% weight by weight (w/w) stannous fluoride (1100 parts per million [ppm] fluoride). Participants then brushed each of the two selected sensitive test teeth first followed by the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
- Sodium Monofluorophosphate: Participants were instructed to dose a dry toothbrush with a full strip (1 inch) of control dentifrice containing 0.76% w/w sodium monofluorophosphate (1000 ppm fluoride). Participants then brushed the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
Period: Overall Study
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Started | 111 | 111
Completed | 111 | 111
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stannous Fluoride: Participants were instructed to dose a dry toothbrush with a full strip (1 inch) of experimental dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride). Participants then brushed each of the two selected sensitive test teeth first followed by the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
- Total: Total of all reporting groups
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate | Total
Number analyzed (Participants) | 111 | 111 | 222
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (10.77) | 47.6 (10.95) | 47.0 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 81 | 163
  Male | 29 | 30 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 109 | 110 | 219
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 15 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 23 | 56
  White | 60 | 73 | 133
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Schiff Sensitivity Score at Baseline [Mean (Standard Deviation); unit: Score on a Scale] — Examiner assessed the participant's response to evaporative air stimulus for each tooth using the Schiff Sensitivity Scale which was scored as follows - 0: Participant does not respond to air stimulation; 1: Participant responded to air stimulus but does not request discontinuation of stimulus; 2: Participant responded to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responded to stimulus, considered stimulus to be painful, and requested discontinuation of the stimulus. A reduction in Schiff Sensitivity score was indicative of an improvement in sensitivity.
  Score on a Scale | 2.50 (0.484) | 2.46 (0.461) | 2.48 (0.472)
Tactile Sensitivity - Tactile Threshold at Baseline [Mean (Standard Deviation); unit: gram (g)] — The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force was reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth.
  gram (g) | 12.66 (4.201) | 13.42 (4.263) | 13.04 (4.240)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score on Day 3
Description: The examiner assessed the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale which was scored as follows - 0: Participant does not respond to air stimulation; 1: Participant responded to air stimulus but does not request discontinuation of stimulus; 2: Participant responded to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responded to stimulus, considered stimulus to be painful, and requested discontinuation of the stimulus. A reduction in Schiff Sensitivity score was indicative of an improvement in sensitivity.
Time Frame: Baseline to Day 3
Population: Analysis for this outcome was performed on intent-to-treat (ITT) population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 111 | 111
Score on a scale | -0.40 (0.485) | 0.00 (0.257)
Statistical Analysis 1: Comparison: Stannous Fluoride vs Sodium Monofluorophosphate; Statistical analyses was conducted under the null hypothesis (H0) of no difference between treatments versus the alternate hypothesis (H1) of a difference between treatments; Test type: Superiority or Other; p < 0.0001, ANCOVA; Change from baseline in Schiff Sensitivity Score as response, treatment as factor and baseline Schiff sensitivity score as a covariate; Least Square (LS) Mean Difference = -0.40, 95% CI 2-sided [-0.505 to -0.300] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favours first named dentifrice

2. Secondary Outcome: Change From Baseline in Tactile Threshold on Day 3
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force was reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth.
Time Frame: Baseline to Day 3
Population: Analysis for this outcome was performed on ITT population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 111 | 111
g | 3.69 (4.941) | 0.09 (2.521)

3. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score Post First Treatment by Direct Application
Description: as for outcome 1
Time Frame: Baseline to 60 seconds post first treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 111 | 111
Score on a scale | -0.17 (0.340) | -0.02 (0.269)

4. Secondary Outcome: Change From Baseline in Tactile Threshold Post First Treatment by Direct Application
Description: as for outcome 2
Time Frame: Baseline to 60 seconds post first treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 111 | 111
g | 1.71 (3.268) | 0.18 (2.328)

ADVERSE EVENTS:
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/111
Other Adverse Events (participants affected / at risk) | 0/111 | 0/111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.